CLINICAL TRIAL: NCT03004495
Title: Open Label, Randomized, Repeated-dose, 3-way Crossover Study to Investigate Pharmacokinetic Interaction and the Safety of Inhaled CHF5259 and CHF6001 Administered in Healthy Subjects Via NEXThaler® Dry Powder Inhaler
Brief Title: Pharmacokinetic Interaction and the Safety of Inhaled CHF5259 and CHF6001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-06302AA1-02
Record Dates: First submitted 2016-10-28; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tanimilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF5259 and CHF6001 (Experimental): (T): CHF6001 + CHF5259 b.i.d. for 14 days
  Interventions: Drug: CHF5259 and CHF6001
- CHF5259 + placebo (Active Comparator): (R1): CHF5259 25µg b.i.d. for 14 days
  Interventions: Drug: CHF5259 + placebo; Other: Placebo
- CHF6001 + placebo (Active Comparator): (R2): CHF6001 b.i.d. for 14 days
  Interventions: Drug: CHF6001 + placebo; Other: Placebo

INTERVENTIONS:
Drug: CHF5259 and CHF6001 — b.i.d. for 14 days
  Other Names: Test Treatment
  Arms: CHF5259 and CHF6001
Drug: CHF5259 + placebo — b.i.d. for 14 days
  Other Names: Reference Treatment 1
  Arms: CHF5259 + placebo
Drug: CHF6001 + placebo — b.i.d. for 14 days
  Other Names: Reference Treatment 2
  Arms: CHF6001 + placebo
Other: Placebo — b.i.d. for 14 days
  Other Names: Matching number of inhalations
  Arms: CHF5259 + placebo; CHF6001 + placebo

SUMMARY:
To evaluate systemic pharmacokinetics of CHF6001 following concomitant administration of CHF6001 and CHF5259, in comparison with the single components, administered in healthy subjects via a multi-dose reservoir NEXThaler® DPI.

DETAILED DESCRIPTION:
This is randomised open label, 3-way cross-over study. Each 14-day treatment period is separated from the following one by a 21-day wash-out period. Subjects will reside at the clinic facilities during the 14 days treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study-related procedure; Healthy males and females volunteers aged 18-55 years inclusive;
* Ability to understand the study procedures and the involved risks, ability to be trained to use the device correctly
* Non smokers or ex-smokers are eligible.
* Good physical and mental status, determined on the basis of the medical history and a general clinical examination;
* Vital signs checked at screening visit and Day -1: Subjects aged 18-45years: Diastolic BP 40-90, Systolic BP 90-140; Subjects aged 46-55 years: Diastolic BP 40-90, Systolic BP 90-150
* 12-lead digitised Electrocardiogram (12-lead ECG) considered as normal (40≤Heart rate≤110bpm,120 ms ≤ PR ≤ 210 ms, QRS ≤ 120 ms, QTcF ≤ 450 ms for males and ≤ 470ms for females) checked at screening;
* Lung function measurements within normal limits: FEV1 > 80% of predicted normal value (according to the Global Lung Function Initiative, ERS Task Force Lung Function Reference Values (1,2) ) and FEV1/FVC ratio > 0.70;
* Male subjects: they and/or their partner of childbearing potential must be willing to use a double contraceptive methods;
* Female subject of non-childbearing potential (WONCBP) Female subjects of childbearing potential (WOCBP) fulfilling one of the following criteria: WOCBP with fertile male partners: they and/or their partner of childbearing potential must be willing to use a double contraceptive methods including one highly effective birth control method and one acceptable birth control method, from the signature of the informed consent and until three months following the last study drug intake; WOCBP with non-fertile male partners: contraception is not required in this case.

Exclusion Criteria:

* Pregnant or lactating women:
* Blood donation (equal or more than 450 ml) or blood loss less than 12 weeks before inhalation of the study medication;
* Positive HIV1 or HIV2 serology; Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C (positive HB surface antigen (HBsAg),HB core antibody ( anti HBc), HC antibody);
* History of substance abuse or drug abuse within 12 months prior to screening visit;
* Clinically significant abnormal 24-h Holter ECG at screening as defined in the Holter interpretative guidelines (Appendix V);
* Any clinically relevant abnormal laboratory value at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment;
* Clinically significant and uncontrolled respiratory, cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, respiratory or psychiatric disorder that may interfere with successful completion of this protocol;
* Subjects with medical diagnosis asthma including childhood asthma;
* Subjects known to have intolerance/ hypersensitivity to M3 Antagonists, or any of the excipients contained in any of the formulations used in the trial;
* Any drug treatment, including prescribed or OTC medicines as well as vitamins, homeopathic remedies etc, taken in the 14 days (3 months for any biologic drugs, enzyme-inducing or enzyme-inhibiting drugs e.g., glucocorticoids, phenobarbital, isoniazid) before the screening visit, with the exception of occasional paracetamol (maximum 2 g per day with a maximum of 10 g per 14 days for mild non-excluding conditions), hormonal contraceptives and hormonal replacement treatment for post-menopausal women;
* Treatment within the previous 3 months before the screening visit with any drug known to have a well defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Plasma CHF 5259 and CHF 6001 AUC 0-12,ss (area under the plasma concentration-time curve from time 0 to 12h post dose at steady on Day 14) | On Day 1 and Day 14 at pre-dose, within 15 minutes from dosing and at the following time points, 5, 10, 15, 30, 45 min and 1, 1.5, 2, 3, 4, 6, 8, 12 h post morning dose. At Day 8, Day 12 and Day 13 at pre-dose
  To evaluate the pharmacokinetic interaction between CHF 5259 and CHF 6001
Plasma CHF 5259 and CHF 6001 Cmax,ss (maximum plasma concentration at steady state on Day 14) | On Day 1 and Day 14 at pre-dose, within 15 minutes from dosing and at the following time points, 5, 10, 15, 30, 45 min and 1, 1.5, 2, 3, 4, 6, 8, 12 h post morning dose. At Day 8, Day 12 and Day 13 at pre-dose
  To evaluate the pharmacokinetic interaction between CHF 5259 and CHF 6001

SECONDARY OUTCOMES:
Plasma CHF 5259 and CHF 6001 and its metabolites (CHF 5956, CHF 6095) AUC0-12h, Cmax, tmax | On Day 1, Day 14 at the following time points: pre-dose, 5, 10, 15, 30, 45 min and 1, 1.5, 2, 3, 4, 6, 8, 12 h post-morning dose.
Holter extracted ECG parameters | On Day 1, Day 14 at the following time points: pre-dose, 5, 10, 15, 30, 45 min and 1, 1.5, 2, 3, 4, 6, 8, 12 h post-morning dose.
Lung function | On Day 1, Day 14: at pre-dose, 5, 15, 30, 45 min and 1, 2 hours post-morning dose
Vital signs | On Day 1, Day 8 and on Day 14 at the following time points: pre-dose, 15 min, 30 min, 1, 2, 4, 8, 12 h post morning dose. From Day 2 to Day 13 at pre-morning dose only, On Day 15 (24 h after last dose), Day 16 (48 h after last dose) and at follow-up. (BP
Plasma CHF 5259 and CHF 6001 and its metabolites (CHF 5956, CHF 6095) Cmax | On Day 1, Day 14 at the following time points: pre-dose, 5, 10, 15, 30, 45 min and 1, 1.5, 2, 3, 4, 6, 8, 12 h post-morning dose.
Plasma CHF 5259 and CHF 6001 and its metabolites (CHF 5956, CHF 6095) tmax | On Day 1, Day 14 at the following time points: pre-dose, 5, 10, 15, 30, 45 min and 1, 1.5, 2, 3, 4, 6, 8, 12 h post-morning dose.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Beboso, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles CPU, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No